CLINICAL TRIAL: NCT07158398
Title: A Phase 1, Open-Label, Fixed-Sequence Study to Evaluate the Effect of Vimseltinib on BCRP and OATP1B1 Inhibition in Healthy Male Participants
Brief Title: Evaluate the Effect of Vimseltinib on the Pharmacokinetics of a BCRP and OATP1B1 Substrate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: DCC-3014-01-007
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rosuvastatin + Vimseltinib (Experimental): Rosuvastatin as single dose will be administered on Day 1 and Day 8. Vimseltinib will be administered every day (QD) on Days 5 through 8.
  Interventions: Drug: Vimseltinib; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Vimseltinib — Administered orally
Drug: Rosuvastatin — Administered orally

SUMMARY:
The main purpose of this study is to determine the effect of Vimseltinib dosing on breast cancer resistance protein (BCRP) and organic-anion-transporting polypeptide 1 B1 (OAT1PB1) activity by using rosuvastatin in healthy male participants. This study will also evaluate the safety and tolerability when vimseltinib is co-administered with rosuvastatin in healthy male participants. This study will last approximately 26 days.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are in good general health, as required by the protocol and as determined by Principal Investigator.
2. Body mass index (BMI) from 18 to 32 kilogram per square meter (kg/m^2).
3. Adequate organ function and blood and urine tests, as required by the protocol and as determined by Principal Investigator.

Exclusion Criteria:

1. History or presence of clinically significant diseases of the neurological, dermatological, renal, hepatic, gastrointestinal, cardiovascular, or musculoskeletal systems or history or presence of clinically significant psychiatric, immunological, endocrine, or metabolic disease as determined by Principal Investigator.
2. Unwilling or unable to comply with the requirements of the protocol.
3. Determined by Principal Investigator to be unsuitable to participate in the study for any other reason.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 20 (Actual)
Dates: Start 2025-10-31 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK): Maximum Observed Plasma Drug Concentration (Cmax) of rosuvastatin | Predose up to 72 hours postdose
PK: Area Under the Concentration Versus Time Curve (AUC) of rosuvastatin | Predose up to 72 hours postdose

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Baseline through Day 26

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team, Study Director — Deciphera Pharmaceuticals, LLC
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No